CLINICAL TRIAL: NCT01944111
Title: Prospective Clinical Trial of Plicated Laparoscopic Adjustable Gastric Banding
Brief Title: Plicated Laparoscopic Adjustable Gastric Banding Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tenet Healthcare Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2315-1
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Weight Loss
Keywords: Gastric plication
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plication (Experimental): Prospective clinical trial comparing Standard Adustable Gastric Banding versus experimental Adjustable Gastric Banding
  Interventions: Device: Plication

INTERVENTIONS:
Device: Plication — Prospective clincial trial comparing adjustable gastric banding with plication versus standard adjustable gastric banding. Variables to be studied include patient age, gender, ethnicity, co-morbid disease conditions, height, weight, BMI, intra-operative data such as operative time and blood loss and post-operative outcomes including length of hosptial stay, complication rates, weight loss, and co-morbid disease resolution.
  Other Names: Lap Band Plication; Adjustable gastric Banding with Plication

SUMMARY:
Compare plicated laparoscopic adjustable gastric banding to standard laparoscopic adjustable gastric banding in prospective clinical trial.

DETAILED DESCRIPTION:
This is a prospective clinical trial comparing experimental plicated adjustable gastric banding versus standard adjustable gastric banding. All enrolled patients will choose to either standard (control group) banding or plication (study group) banding. Each patient will complete a standardized survey rating their satisfaction from surgery, their satiety levels and Green Zone Patient Questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Morbidly Obese
* BMI >40 or
* BMI >35 plus co-morbid obesity related disease conditions
* Without contraindications to bariatric surgery: eg pregnancy, desire to become pregnant within the next 12 months, myocardial infarct within the last 6 months, cancer within last 5 years, end stage renal/liver disease
* Without any metabolic or medically correctable causes for obesity: eg untreated hypothyroidism, Prader-Willi

Exclusion Criteria:

* Any patient not meeting the inclusion criteria
* Patients with any major medical problems contraindicating surgery
* Patients with a medically treatable cause of obesity
* Patients who elect to undergo a surgery other than Plication adjustable gastric banding or standard adjustable gastric banding
* Alcohol or drug addiction
* Established infection anywhere in the body at the time of surgery
* Previous history of bariatric surgery, intestinal obstruction, or adhesive peritonitis
* Family or patient history of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Weight loss | at least 1 year
  Weight loss 4 weeks post surgical:20% additional than without plication, 3months post surgical: 30% additional than without plication, 6 months post surgical:30-40% additional than without plication, 1 year post surgical = 30-40% additional than without plication & at 1 year patient will require 50% fewer adjustments than without plication.

CONTACTS AND LOCATIONS:
Overall Officials: James S Scott, MD, Principal Investigator — Tenet Healthcare Corporation
Locations (1):
- Des Peres Hospital, St Louis, Missouri, United States